CLINICAL TRIAL: NCT06816108
Title: A Phase I, Open-label, Dose Escalation Study to Evaluate the Tolerability and Safety of ONO-7428 in Participants With Unresectable Advanced or Recurrent Solid Tumors
Brief Title: A Study of ONO-7428 in Participants With Unresectable Advanced or Recurrent Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7428-01
Record Dates: First submitted 2025-01-29; First posted 2025-02-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor; NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONO-7428 (Experimental)
  Interventions: Drug: ONO-7428

INTERVENTIONS:
Drug: ONO-7428 — Specified dose on specified days

SUMMARY:
This study is to evaluate the tolerability and safety of ONO-7428 in participants with unresectable advanced or recurrent solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with histologically or cytologically confirmed unresectable advanced or recurrent solid tumors.

   [Backfill cohort only] Participants with histologically or cytologically confirmed Stage IIIB, IIIC, IV, or recurrent NSCLC according to UICC-TNM classification.
2. Participants who are refractory or intolerant to standard therapy.
3. Participants with a tumor type for which anti-PD-(L)1 antibodies have been approved and who have previously treated with anti-PD-(L)1 antibody containing regimen.
4. Participants with Eastern Cooperative Oncology Group Performance Status 0 or 1.
5. Participants with tumor tissue samples available for biomarker testing.

Exclusion Criteria:

1. Participants with a complication or history of severe hypersensitivity to any other antibody drugs.
2. Participants with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease
3. Participants with severe peritoneal dissemination.
4. Participants with pericardial fluid, pleural effusion, or ascites requiring treatment.
5. Participants with uncontrolled tumor-related pain.
6. Participants with active or history of interstitial lung disease or pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities（DLT） | 21 days
Adverse event (AE) | Up to 2 years

SECONDARY OUTCOMES:
Cmax | Up to 2 years
Tmax | Up to 2 years
Area under the Plasma Concentration versus Time Curve (AUC) | Up to 2 years
Ctrough | Up to 2 years
Objective Response Rate (ORR) | Up to 2 years
Disease Control Rate (DCR) | Up to 2 years
Overall Survival (OS) | Up to 2 years
Progression-Free Survival (PFS) | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Time to Response (TTR) | Up to 2 years
Best Overall Response (BOR) | Up to 2 years
Percent change from baseline in the sum of diameters of target lesions | Up to 2 years
Best reduction percent change from baseline in the sum of diameters of target lesions | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (15):
- Japan (15):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Kyoto University Hospital, Kyoto, Kyoto
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Saitama Cancer Center, Shinden, Saitama
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō-Ku, Tokyo
  - The Cancer Institute Hospital Of JFCR, Koto-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No